CLINICAL TRIAL: NCT00494611
Title: A Study of the Perioperative Use of Cetuximab in Colon Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit subjects in timely fashion for the study
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Dr. Richard Whelan, St Luke's Roosevelt Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAC3683
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-06

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Peri operative Cetuximab. — Cetuximab will be given immediately preoperative and early post surgery period.
  Other Names: Cetuximab (IMC-C225-marketed under the name Erbitux)

SUMMARY:
There are more than 140,000 new cases of colon cancer diagnosed each year, and over 60,000 Americans die from colon cancer annually. To date, surgical resection remains the mainstay of treatment for colon cancer. However, between 35% and 45% of patients, despite colon surgery, retain unseen tumor cells in the bloodstream or in small clumps in the liver or other tissues. It is for this reason that postoperative chemotherapy (anti-tumor drugs) is recommended and given to some patients after surgery. Conventional chemotherapy is usually started no earlier than 4 to 6 weeks after the colon cancer has been resected.

Despite surgery and conventional chemotherapy, a significant number of patients develop cancer recurrences and many go on to die from the cancer. For this reason, investigators continue to look for new cancer treatments and approaches. The study under consideration proposes to give colon cancer patients an anti-cancer therapy for 3 weeks before and for 3 weeks after undergoing operation to remove the colon cancer. This time period is referred to as the "perioperative period." Presently, around the world, doctors do not administer any type of anti-cancer therapy during the perioperative period. It is the belief of the investigators carrying out this study that this period may be an ideal time to fight the tumor and that treatment given during this time may improve survival and reduce cancer recurrence rates. Patients who choose to receive this biologic anti-cancer treatment immediately before and after surgery can also receive conventional chemotherapy at the usual time (4-6 weeks after surgery). Thus, this perioperative anti-cancer treatment would not interfere with the standard chemotherapy regimens used today.

The drug that is to be given in this study is called Cetuximab (also known as "Erbitux"). This is an anti-cancer drug which has already been approved by the FDA for use in patients who have colon cancer. This drug, like all of the other anti-cancer drugs used for treating colon cancer, has been given either well after surgery or to patients with very advanced disease who have not undergo surgery. What is unique about the St. Luke's Roosevelt study is that the drug will be given during the 3 weeks before surgery and for the first 3 weeks after the colon resection surgery.

To summarize, Cetuximab is a humanized antibody to EGFR which has been shown to be effective in killing tumor cells in patients with colon cancer.

In this study the Cetuximab is to be given 1) after the surgery, 2) immediately before the operation, or 3) both before and after surgery. Entry into the study means that the operation may be delayed for at least 3 weeks in order for the drug to be given. Since many patients who do not participate in any research studies wait at least that long for surgery this does not constitute a delay. The drug has a safety profile and has been well tolerated, in general. However, since thus far it has not been given in the weeks immediately prior to or immediately after major surgery there is no safety profile for this drug during the perioperative period. The primary goals of this preliminary study are to establish the safety of Cetuximab in the perioperative period and to demonstrate that the preoperative doses have an actual impact on the tumor cells themselves.

DETAILED DESCRIPTION:
Cetuximab's tumor growth inhibitory mechanism directly blocks EGFR. After binding to EGFR, the antibody blocks signal transduction through the receptor with a subsequent inhibition of tumor cell proliferation and MMP expression. We hypothesize that peri-operative weekly administration of Cetuximab, a humanized monoclonal antibody to EGF receptor (EGFR), for 3 weeks immediately prior to surgery and for 3 weeks immediately after colon cancer surgery is safe. This drug has been demonstrated to be effective in Stage 4 colon cancer patients and is approved for use in colorectal cancer patients. Cetuximab has never been administered in the month immediately before or after colon surgery. Establishing the safety of Cetuximab in the perioperative setting is the primary objective of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 18 and 85 years of age and have biopsy proven adenocarcinoma of the large bowel at least 2 cm in size.
* Patients receiving preoperative study drug will not have undergone operation with resection and pathologic staging and so will be Stage 1 or 2 or 3 patients. Patients in groups who only receive postoperative study drug will be Stage 3 patients only.
* Patients may be of any race and either gender.
* Patients without evidence of Stage 4 cancer on the basis of preoperative chest X-rays, abdominal and pelvic CT scans (preferably with IV and oral contrast), or other metastatic work up (USG, PET, MRI) will be eligible for entry.
* Only those patients with colon tumors located between the proximal rectum (defined as 15 cm from the anal verge) and the cecum who are to undergo elective resection will be eligible for this study.
* Those patients with a reasonable performance status (ECOG Performance Status Scale score of O or 1) will be eligible for entry into the study.
* Those patients whose renal, hepatic, and hematologic blood test values meet the following criteria will be eligible (as per the Columbia Presbyterian clinical chemistry lab):

  * Hemoglobin >8.0g/dL
  * Neutrophils >1.5 x 10^9/L
  * Lymphocytes >1.2 x 10^9/L
  * Platelets >100 x 10^9/L
  * Serum creatinine <1.8 mg/dL
  * Serum bilirubin <2mg/dL
  * SGOT <41mg/dL
  * SGPT <41mg/dL

Exclusion Criteria:

* Patients with tumors less than 2 cm in size or those with polyp cancers that have been fully removed or those who have had partial removal endoscopically where the remnant is less than 2 cm in size are not eligible.
* Patients with a history of a second current malignancy or past malignancy (within the past 5 years), other than the colon neoplasm in question (excepting basal cell skin carcinomas) will not be eligible for entry into this study.
* Patients with rectal cancer (located between the anus and 15 cm proximal to the anal verge) or Stage 4 colon cancer are not eligible.
* Patients with a history of immunosuppression secondary to a disease process, current steroid usage, or the use of other immunosuppressive drugs, within three months of the planned surgery, will not be eligible for this study.
* Patients with Hepatitis B or C or who are HIV positive will be excluded.
* Patients who have received chemotherapy or radiotherapy within 3 months of the anticipated surgery will not be eligible.
* Patients with bowel obstruction, or other emergency indications for surgery, will not be eligible.
* Pregnant or nursing patients are not eligible for entry into the study.

  * All WOCBP must have a negative pregnancy test within 7 days prior to first receiving investigational product. If the pregnancy test is positive, the patient will not receive cetuximab and will not be eligible for entry into the study.
  * In addition, all WOCBP will be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
  * Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors associated with an unintentional pregnancy in this setting. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.)
  * The Investigator will immediately notify both the IRB and Bristol Meyers Squibb in the event of a confirmed pregnancy in a patient participating in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety of peri operative Cetuximab. | within 90 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Whelan, MD, Study Chair — Columbia University
Locations (1):
- St Luke's Roosevelt Medical Center, New York, New York, United States